CLINICAL TRIAL: NCT00110344
Title: A Phase II Study of BAY 43-9006 Prior to and Following Nephrectomy in Patients With Metastatic Renal Cell Carcinoma.
Brief Title: Research Study for Patients With Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11547
Record Dates: First submitted 2005-05-06; First posted 2005-05-09 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Carcinoma, Renal Cell
Keywords: Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — Cycle 1. Patients are randomized in a double-blind fashion to receive either Nexavar (Sorafenib, BAY 43-906; this arm) or matching placebo (see below) for 14 days. Dose range will be depending on hematologic and other toxicity between 400 mg (2 tablets of 200 mg) orally twice bid and 400 mg orally every 2 days. Cycle 2: patients who are eligible undergo nephrectomy. After the post-nephrectomy recovery period, all patients will receive 400 mg of BAY 43-906, twice daily (administered as two 200 mg tablets) in an open-label fashion.Cycle 3+: 400 mg of BAY 43-906, twice daily (administered as two 200 mg tablets) in an open-label fashion.
  Arms: Arm 1
Drug: Placebo — Cycle 1. Patients are randomized in a double-blind fashion to receive either Nexavar (see above) or matching placebo (this arm) for 14 days. Dose range will be depending on hematologic and other toxicity between 400mg (2 tablets of 200mg) orally twice bid and 400mg orally every 2 days. Cycle 2 and 3: see above (no placebo application)
  Arms: Arm 2

SUMMARY:
This study has been designed to study patients diagnosed with advanced renal cell cancer with the primary tumor in place.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Clinical, radiographic, or pathologic diagnosis of metastatic renal cell carcinoma (RCC). All renal cell histologies are allowed- Acceptable surgical risk in the judgment of the study investigator and consulting urological surgeon
* At least one uni-dimensional measurable lesion outside the planned nephrectomy specimen
* Patients who have an ECOG performance status of 0 or 1 Exclusion Criteria:
* History of bleeding diathesis or unexpected surgical bleeding- Patients currently receiving treatment with or having a requirement for therapeutic anticoagulation
* Prior therapy for RCC. Palliative radiation therapy for painful or unstable bone metastases is permitted provided that there is measurable metastatic disease outside the radiation field
* Known history of HIV infection- Symptomatic metastatic brain or meningeal tumors, unless the patient is > 6 months from definitive therapy, has a CT or MRI scan within 6 weeks of study entry negative for brain metastases and is clinically stable with respect to the tumor at the time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-11; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Best Overall Response Rate (complete and partial response rate) | During study treatment or within 30 days after termination of active therapy

SECONDARY OUTCOMES:
Progression-free survival | Last date of tumor assessment
Overall response rate | Last day of tumor assessement
Time to response | throughout study
Safety | all visits

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Boston, Massachusetts, United States